CLINICAL TRIAL: NCT04551209
Title: "Effect Of Apical Patency On Post-Operative Pain After Single Visit Endodontic Treatment In Necrotic Teeth With Asymptomatic Apical Periodontitis: A Quasi Experimental Study"
Brief Title: "Effect of Apical Patency on Post-endodontic Pain"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Medical Sciences, Pakistan (Other)
Responsible Party: Principal Investigator, Yousaf, Assistant Professor / Consultant, National University of Medical Sciences, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 905/Trg-ABP1K2
Record Dates: First submitted 2020-07-24; First posted 2020-09-16 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Apical Periodontitis
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apical patency group (Experimental): Patients in which apical patency is maintained.
  Interventions: Procedure: Maintaining apical patency
- Non- apical patency group (No Intervention): Patients in which apical patency is not maintained

INTERVENTIONS:
Procedure: Maintaining apical patency — In apical patency group, a size 10 K file will be passed beyond the apical foramen between each instrument change to maintain apical patency while in Non apical patency group, K file will be carried up to the working length only. A final peri-apical radiograph will be taken in the group A with the 10 K patency file 01mm beyond the apical foramen to confirm patency.
  Arms: Apical patency group

SUMMARY:
This study is designed to find out the effect of maintaining apical patency versus non maintaining apical patency on post-operative pain after single visit endodontic treatment in necrotic teeth with asymptomatic apical periodontitis

DETAILED DESCRIPTION:
After taking approval from the ethical committee (AFID No 905/Trg-ABP1K2), this study is planned at operative department in Armed Forces Institute of Dentistry, Rawalpindi from 01 June 2020 to 31 December 2020. Informed consent would be taken from 240 patients of 20-50 years of age from both gender with good general, mental and physical health who would be selected for this study and would be randomly divided into two equal groups with the help of scientific random number table.

The mandibular first molar teeth with asymptomatic apical periodontitis either with necrotic pulps, without any intra-oral or extra-oral swelling or any draining sinus tract will be selected for this study. Patients on preoperative analgesics and antibiotics, teeth with calcified canals and open apex, previously traumatized teeth and root canal treated teeth along with immune-compromised patients, pregnant and lactating mothers will be excluded from this study.

The patients reporting to the Operative Dentistry Department of Armed Forces Institute of Dentistry, Rawalpindi requiring root canals of their mandibular first molar will be screened for inclusion by taking history, performing relevant clinical examination and necessary investigations along with peri-apical radiographs. The whole procedure of the study will be explained to the patients in Urdu. After taking written informed consent from the willing participants of this study the procedure will be started. Two groups will be formed:

Group A: Patency group and Group B: Non-patency group Root canal treatment will be initiated under local anesthesia and rubber dam isolation. Working length will be taken with apex locator and will be confirmed with radiograph. The root canals will be instrumented with ProTaper Next system under copious irrigation with 5.25% sodium hypochlorite (NaOCl) and 17% EDTA solution.

In group A, a size 10 K file will be passed beyond the apical foramen between each instrument change to maintain apical patency while in group B, K file will be carried up to the working length only. A final peri-apical radiograph will be taken in the group A with the 10 K patency file 01mm beyond the apical foramen to confirm patency.

To control the microbiological impact on post-operative pain 2.5% sodium hypochlorite and 17% EDTA will be used as irrigants in both groups. Obturation will be done with cold lateral condensation using Pro Taper Next GP points and permanent restoration will be done with composite. At the end of this appointment patients will be given a visual analogue scale (VAS), and will be advised to mark at the scale according to his pain intensity after 24 hours and 48 hours after the treatment and will be asked to bring these reading with him on the next scheduled visit after one week for tooth preparation for metal ceramic crown. Patients will be given analgesic and will be advised to take it only in case of severe pain. VAS scores of less than 4 will be considered as no pain, score of 4-7 will be considered as mild and/or moderate pain and scores of 8 and above will be considered as severe pain. (no pain = <3, moderate pain = >4 to 7, severe pain = > 8). Frequencies, percentages, mean and standard deviation will be calculated for qualitative variable like inter appointment pain and for quantitative variables like gender; mean and standard deviation along with percentages in each group will be calculated with SPSS 22. Chi-square test will be used to compare the frequency of pain between the two groups after 24 and 48 hours of endodontic treatment. The p value of <0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Necrotic Mandibular first molar teeth with asymptomatic apical periodontitis
* Mandibular first molar teeth without any intra-oral or extra-oral swelling or any draining sinus

Exclusion Criteria:

* Patients on preoperative analgesics and antibiotics
* Mandibular first molars with calcified canals and open apex
* Previously traumatized teeth and root canal treated teeth
* Immune-compromised patients
* pregnant and lactating mothers

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Post operative pain as determined by VAS (Visual Analogue Scale) | 06 months
  To find out the incidence of post operative pain with Visual analogue scale after single visit endodontic treatment in necrotic teeth with asymptomatic apical periodontitis in two groups, Group A of 120 patients in which apical patency is maintained and Group B of 120 patients in which apical patency is non maintained. VAS (Visual Analogue Scale) will be used to measure pain. VAS scores of less than 4 will be considered as no pain, score of 4-7 will be considered as mild and/or moderate pain and scores of 8 and above will be considered as severe pain. (no pain = <3, moderate pain = >4 to 7, severe pain = > 8).

CONTACTS AND LOCATIONS:
Overall Officials: Dil Rasheed, Study Director — AFID
Locations (1):
- Afid, Nums, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No